CLINICAL TRIAL: NCT06731036
Title: A Compassionate Release Protocol: Expanded Access to CD34+ Selection Utilizing Miltenyi CliniMACS Prodigy® for Patients Receiving Peripheral Blood Stem Cell Transplantations and Stem Cell Boosts
Brief Title: Expanded Access to CD34+ Selection Utilizing Miltenyi CliniMACS Prodigy® for Patients Receiving Peripheral Blood Stem Cell Transplantations and Stem Cell Boosts
Status: Available | Type: Expanded Access
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UF-PEDS036; IRB202401729 (Other: University of Florida)
Record Dates: First submitted 2024-12-04; First posted 2024-12-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Severe Combined Immunodeficiency; Fanconi Anemia; Dyskeratosis Congenita; Sickle Cell Disease
Keywords: stem cell transplantation; graft manipulation
MeSH Terms: conditions — Severe Combined Immunodeficiency; Fanconi Anemia; Dyskeratosis Congenita; Anemia, Sickle Cell

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: CD34+ cell enriched stem cell graft — Patients will receive a peripheral blood stem cell graft that has been CD34+ cell enriched using the Miltenyi CliniMACS Prodigy® system.

SUMMARY:
Allogeneic stem cell transplantation (alloSCT) is utilized for various underlying diseases. AlloSCT is limited by graft versus host disease (GVHD), graft rejection, viral infections, and post-transplant lymphoproliferative disorders. To mitigate graft versus host disease, graft manipulation has been taking place with CD34+ selection to decrease T-cells entering into the patient, thus lowering the risk of GVHD.

Historically CD34+ manipulation has been performed under a humanitarian use device by utilizing the Miltenyi CliniMACs CD34 Reagent System. This was used for patients with AML in first remission. This approach has additionally been used for patients with sickle cell disease, immune deficiencies, and poor graft function with excellent efficiency. The purpose of this protocol is to create expanded access of CD34+ manipulation for various underlying diseases utilizing the Miltenyi CliniMACS Prodigy® device.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 1 month of age
* The following category of patients is eligible for this protocol:

  a. Patients undergoing allogeneic transplantation for the following indications:

  i. Non-malignant disorders where graft versus host disease is detrimental:
* Severe combined immune deficiency
* Fanconi Anemia
* Dyskeratosis Congenita
* Sickle Cell Disease

or

b. Patients undergoing autologous transplantation intended for hematopoietic/immunologic reconstitution

or

c. Patients with poor graft function defined as persistent cytopenia following stem cell transplant without evidence of recurrent disease

* Subjects must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician and approved by the PI] may be included).
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout participation at least 1 year after the stem cell infusion to minimize the risk of pregnancy. Prior to protocol enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. WOCBP includes any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:

  1. Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or
  2. For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.

     * Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout participation and should avoid conceiving children for 1 year following infusion of the stem cells.

Exclusion Criteria:

* Patients with a fully HLA matched sibling donor
* Patients with active graft versus host disease
* Patient with uncontrollable transplant associated thrombotic microangiopathy
* Patient not cleared by transplant provider to process
* Donor unable to donate peripheral blood stem cells
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire participation period and for at least 1 year after stem cell infusion.
* Females who are known to be pregnant or breastfeeding.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 1 Month | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Milner, MD, Principal Investigator — University of Florida